CLINICAL TRIAL: NCT04385680
Title: The Impact of Chlorhexidine Preoperative Vaginal Preparation in Reducing the Post-cesarean Endometritis and Sepsis for Cases in Labor. A Randomized Controlled Trial
Brief Title: Chlorhexidine Vaginal Preparation for Reduction of Post-cesarean Endometritis and Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate Professor Obstetrics & Gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: chlorhex. post cs endometritis
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Postpartum Endometritis; Wound Infection; Chlorhexidine Adverse Reaction; Postoperative Fever
Keywords: post-cesarean endometritis; wound infection; chlorhexidine vaginal preparation; chlorhexidine adverse reaction
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine vaginal prep.arm (Experimental): Women in labor who will receive vaginal cleaning immediately before cesarean section using 50 ml of chlorhexidine gluconate 0.05% solution and standard abdominal scrub with chlorhexidine gluconate 4%. This concentration is indicated within the British National Formulary for swabbing in obstetrics. A swab soaked in the antiseptic will be used to clean the vagina for 30 seconds prior to CS at the time of urinary catheter insertion by long forceps.
  After the CS procedure, the vagina is always cleaned of excess blood as with a dry swab.
  Interventions: Drug: Chlorhexidine Gluconate vaginal solution 0.05%
- No vaginal antiseptic arm (No Intervention): Women in labor who will receive abdominal scrub with chlorhexidine gluconate 4% only. Vaginal preparation is not including antiseptic or using normal saline only.

INTERVENTIONS:
Drug: Chlorhexidine Gluconate vaginal solution 0.05% — preoperative vaginal preparation
  Other Names: No preparation or preparation with saline only
  Arms: Chlorhexidine vaginal prep.arm

SUMMARY:
The study aims to assess the beneficial value of vaginal preparation with chlorhexidine gluconate 0.05% before cesarean delivery of cases in labor in reduction of postoperative endometritis, fever and wound complications compared to no preparation or using saline only.

DETAILED DESCRIPTION:
Despite the demonstrated effectiveness of the vaginal cleansing in the previous study, yet this has not been adopted within obstetric practice internationally and does not feature within the NICE Intrapartum guideline.7 This is may be due to concerns with exposure of the fetus to iodine-based substances, concerns with vaginal staining and allergy to iodine. Iodine is an antibacterial agent, but becomes inactive by the presence of blood may limit its use.

Chlorhexidine show greater reduction in skin flora after application compared with povidone-iodine agents (0.5 and 4%) respectively and has a greater residual activity after application than other preparations and (unlike povidone iodine) it is not inactivated by the presence of blood. Thus, there are a number of reasons to believe that vaginal cleansing with chlorhexidine would be an appropriate alternative to povidone iodine.8 There is one RCT comparing povidone iodine with chlorhexidine gluconate for vaginal cleansing at CS. This suggested that chlorhexidine may be superior, and further research was needed.9 Solutions that contain lower concentrations, such as chlorhexidine gluconate and acetate (0.05%) are usually well tolerated and may be used for vaginal preparation. With this preparation, there are no reported cases of allergy.8 Importantly, no safety concerns for the mother or baby have been identified with chlorhexidine gluconate used for vaginal cleansing.10

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥28 weeks.
2. Cases had cesarean section after start of labor.

Exclusion Criteria:

1. Women with known allergy to chlorhexidine gluconate or any of its ingredients.
2. Women with diagnosed group B streptococcus (GBS) colonization.
3. Women with active infection during the procedure.
4. Women did not receive the standard preoperative antibiotic prophylaxis.
5. Women with diagnosis of chorioamnionitis.
6. Prolonged rupture of membranes >7 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
post-cesarean endometritis | First 10 days post-cesarean
  uterine fundal tenderness on bimanual examination ( physical examination: suprapubic tenderness, pain elicited by cervical motion, tenderness in parametrium, all during bimanual examination) + with fever (An oral temperature of 38°C or higher within the first 10 days postpartum or 38.7°C within the first 24 hours postpartum) ± purulent lochia requiring antibiotic therapy ( initial antibiotic will be started then waiting for proper therapy according to culture and sensitivity
Postoperative wound infection | First month after cesarean
  erythema, warmth, tenderness, purulent drainage from the incision site, with or without fever, requiring antibiotic therapy.

SECONDARY OUTCOMES:
Significant leukocytosis | First 10 days postcesarean
  increase of WBCs count > 50% from preoperative count
Chlorhexidine adverse drug reaction | First 10 days
  maternal or neonatal allergy or irritation
incidence of hospital readmission | One month
  percent of cases needed readmission in both arms
length of hospital stay | One month
  duration of hospitalization due to endometritis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shafiek, Principal Investigator — Armed forces hospitals Southern Region KSA; Hytham Atia, Principal Investigator — Armed Forces Hospitals Southern Region
Locations (1):
- Armed Forces Hospitals Southern Region, Khamis Mushait, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256
- [Background] Haas DM, Morgan S, Contreras K, Enders S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2018 Jul 17;7(7):CD007892. doi: 10.1002/14651858.CD007892.pub6. PMID 30016540